CLINICAL TRIAL: NCT04907565
Title: Impact of Obesity on Post-operative Cognitive Dysfunction: Role of Adipose Tissue
Acronym: ODCOTA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0014
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Cognitive Impairment; Post-Operative Confusion
Keywords: Obesity; Post-operative cognitive dysfunction; Inflammation; Inflammatory cytokines
MeSH Terms: conditions — Obesity; Cognitive Dysfunction; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and white adipose tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Obese patients: BMI >30kg/m2
  Interventions: Biological: Blood sampling; Biological: white adipose tissue sampling
- non obese patients: BMI between 18 to 29kg/m2
  Interventions: Biological: Blood sampling; Biological: white adipose tissue sampling

INTERVENTIONS:
Biological: Blood sampling — 4 tubes of 7 mL of blood will be collected
Biological: white adipose tissue sampling — At the beginning of the surgery, samples of white adipose tissue from the surgical wound will be collected.

SUMMARY:
This research aims at describing the relationship between white adipose tissue inflammation and post-operative cognitive dysfunctions.The possible link between inflammatory cytokines secretions of the white adipose tissue of a surgical wound and the arising of patient's cognitive dysfunction in the post-operative course will be investigated. The hypothesis is that obese patient's inflammation of the white adipose tissue leads to cognitive dysfunction.

DETAILED DESCRIPTION:
The postoperative cognitive dysfunctions (POCD) are characterized by delirium and cognitive impairment. The delirium is defined by an acute altered attention with a fluctuating course. The post-operative cognitive impairment involves the early alteration of different functions including memory, attention and cognitive flexibility. POCD have a major impact in patient's morbidity. They are linked to the systemic inflammation induced by the surgical wound. The systemic inflammation leads to the rupture of the brain-blood barrier and to hippocampal inflammation. As hippocampus mediates the principal cognitive functions, hippocampal inflammation leads to POCD. Orthopedic and cardiac surgery are particularly concerned. Obesity is growing condition in the French population. It is linked to chronic systemic inflammation and altered cognitive functions. We think that obese people may present a susceptibility to POCD because of the pre-operative systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* patient about to receive a hip arthroplasty under general anesthesia, elective cardiac surgery with cardiopulmonary bypass,
* patient with a MMSE score > or = 20(/30),
* patient able to give informed consent

Exclusion Criteria:

* emergency surgery, or surgery in a septic context,
* patient with a known dementia or altered MMSE score (under 20)

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prospective, monocentric study conduct in Toulouse university hospital
Sampling Method: Probability Sample
Enrollment: 408 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2025-09-21 (Estimated)

PRIMARY OUTCOMES:
Arising of POCD measured by a composite criterion | day 5 after surgery
  2 points Mini-Mental State Examination (MMSE) score decrease compared to the pre-operative score, and/or appearance of a delirium tracked down every day by the Confusion Assessment Method (CAM) during the hospital course.

SECONDARY OUTCOMES:
Variation of inflammatory cytokine levels from patient's plasma and patient's white adipose tissue (extract from a controlled medium). | Day 0 and day 5 after surgery
  inflammatory cytokine levels will be measured in plasma and adipose tissue, and compared.
Identification of a linked between inflammatory cytokine levels and the appearance of POCD. | day 5 after surgery
  inflammatory cytokine levels will be measured in plasma and adipose tissue, and correlated with appearance of POCD
Peri-operative variations of the protein S100B, an autonomy scale (IADL) and a quality of life scale (EQ5D). | day 5 after surgery
  protein S100B levels will be measured in plasma and adipose tissue, and correlated with scores of autonomy scale (IADL) and quality of life scale (EQ5D).

CONTACTS AND LOCATIONS:
Overall Officials: François Labaste, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Purpan University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No